CLINICAL TRIAL: NCT05498090
Title: Interrogating Fatty Acid Metabolism Impairment and Clinical Correlates in Males with Klinefelter Syndrome
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-2860
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-04

CONDITIONS: Klinefelter Syndrome
Keywords: Klinefelters; XXY; 47, XXY; Klinefelter's Syndrome; Klinefelter
MeSH Terms: conditions — Klinefelter Syndrome | interventions — Fenofibrate

STUDY DESIGN:
Intervention Model Description: 2 arms in study: cross-sectional (cases v. controls); interventional (cases only: pre and post fenofibrate intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Cross-sectional, Cases v. Controls) (No Intervention): Cases (those with Klinefelter) vs. controls (those without Klinefelter)
- Arm 2 (Interventional with cases) (Experimental): Cases (those with Klinefelter); Comparison of outcomes pre and post fenofibrate intervention, 145mg PO daily for 4 weeks
  Interventions: Drug: Fenofibrate 145 mg

INTERVENTIONS:
Drug: Fenofibrate 145 mg — Fenofibrate 145 mg PO daily for 4 weeks
  Arms: Arm 2 (Interventional with cases)

SUMMARY:
This study will learn more about how the body uses energy. Usually, the body uses sugars as energy first and then fats are used when the sugar stores are gone. Some people have trouble using fats as energy. This can lead to feeling tired, difficulty exercising, and storing too much fat where it does not belong (like in the muscle). It is believed that some boys and men with Klinefelter Syndrome may not be able to use fats as energy normally, and that a medication called fenofibrate could help this.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Ages 15 to 40 years
* Total testosterone concentration within the normal range for age and pubertal stage
* For the KS group only: genetic testing results confirming KS

Exclusion Criteria:

* Liver disease (ALT or AST > 3x upper limit of normal)
* Renal impairment (estimated creatinine clearance <80 ml/min)
* Diabetes mellitus (A1c > 6.4%)
* Untreated hypogonadism
* Treatment with a PPAR agonist (including fish oil) or statin within the past month
* Unstable medications with any medication added or removed within the past 2 weeks or plan for medication changes during the study period
* Inability to tolerate study procedures, including any medical conditions that make exercise unsafe at the discretion of the study physician
* For the KS group only: known allergy to fibrates, inability to swallow tablets

Ages: 15 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
maximal rate of fat oxidation | 1 month
  maximal rate of fat oxidation during prolong submaximal exercise
skeletal muscle fat oxidation | 1 month
  Maximal skeletal muscle mitochondrial respiration with lipid substrate

SECONDARY OUTCOMES:
differentially-expressed genes in plasma | 1 month
  Expression levels of UCP2, PLTP, CRAT, ECH1, SLC27A1, SLC27A4, CPT1B from fasting blood draw
differentially-expressed genes in skeletal muscle tissue | 1 month
  Expression levels of UCP2, PLTP, CRAT, ECH1, SLC27A1, SLC27A4, CPT1B from skeletal muscle biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Shanlee M Davis, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States